CLINICAL TRIAL: NCT07158125
Title: Role of Th17 and Stress-related Neuroendocrine Markers in the Pathogenesis of Periodontal Disease in Individuals With Psoriasis
Brief Title: Pathogenesis of Periodontal Disease in Individuals With Psoriasis
Status: Not yet recruiting | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Dilek KARADOĞAN, Assoc. Prof. Dr., Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: periopsoriasis06/2025
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Psoriasis
Keywords: psoriasis; periodontitis; Th17; cortisol; dehydroepiandrosterone; chromogranin A
MeSH Terms: conditions — Psoriasis; Periodontitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Gingival Crevicular Fluid (GCF) Collection Samples will be collected from four different teeth from each participant, each with the deepest pocket. After isolating the teeth, paper strips will be carefully placed in the sulcus; the strips will be left in the sulcus/pocket for 30 seconds. The GCF volume of each strip will be measured using a pre-calibrated electronic device (Peritron 8000).
  Saliva Sampling Participants will be asked to rinse their mouths with water and wait 5 minutes to prevent contamination. After waiting, they will be asked to collect saliva in the bottom of their mouths and then spit into a sterile metal cup for another 5 minutes. Unstimulated saliva samples will be transferred to sterile Eppendorf tubes. Saliva flow rate will be calculated by dividing the total saliva volume by the collection time for each participant.
  Samples will be stored at -80°C until the day of laboratory analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- No psoriasis severity: Patients with a PASI (Psoriasis Area and Severity Index) score of 0
- Mild psoriasis severity: Patients with a PASI (Psoriasis Area and Severity Index) score of 1-10
- Moderate psoriasis severity: Patients with a PASI (Psoriasis Area and Severity Index) score of 10-20
- Severe psoriasis: Patients with a PASI (Psoriasis Area and Severity Index) score of >20

SUMMARY:
The aim of this study is to evaluate the levels of Th17 cell-associated cytokines (IL-17, IL-21, IL-23) and the salivary stress biomarkers cortisol, dehydroepiandrosterone, and Chromogranin A in the pathogenesis of periodontal disease in individuals with psoriasis, thereby revealing immunological and neuroendocrine interactions.

The fundamental question it aims to answer is:

What are the biological mechanisms that may increase the risk of periodontal disease in individuals with psoriasis?

In this context, the periodontal status of individuals with psoriasis will be clinically assessed, followed by analysis of the levels of Th17-associated cytokines and stress biomarkers in gingival crevicular fluid and saliva samples. Additionally, patients will be asked questions from the Social Appearance Anxiety Scale. The periodontal status of individuals with psoriasis will be determined cross-sectionally, and the resulting biomarker levels will be examined. In addition, the data obtained will be evaluated with statistical analysis in relation to disease severity and clinical parameters.

DETAILED DESCRIPTION:
Psoriasis and periodontitis are chronic inflammatory diseases, and Th17 cells and their secreted cytokines, such as IL-17, IL-21, and IL-23, have been shown to play a significant role in the pathogenesis of both. Recent studies suggest a possible immunological link between these two diseases. Furthermore, in a stress-induced disease like psoriasis, the effects of chronic stress on the immune system are attracting increasing attention. The interaction of neuroendocrine markers, such as cortisol, dehydroepiandrosterone (DHEA), and chromogranin A (CgA), released via the hypothalamic-pituitary-adrenal axis, with immune responses and inflammatory processes may play a significant role in the development of periodontal disease.

This project will jointly examine the immunological and neuroendocrine basis of periodontal disease in individuals with psoriasis. Cortisol, DHEA, and CgA levels will be measured in saliva samples, and the relationship between these biomarkers and periodontal parameters will be analyzed. Cytokine levels related to the Th17 pathways will be examined in gingival crevicular fluid to reveal the impact of psoriasis on periodontal tissue. The Social Appearance Anxiety Scale will also be administered. All data obtained will be statistically analyzed.

In this context, this study aims to investigate the role of these two chronic and inflammatory diseases (periodontitis and psoriasis) in the Th17 axis based on stress biomarkers (IL-17, IL-21, and IL-23). Thus, we plan to evaluate the relationship between periodontitis and psoriasis biochemically using salivary stress markers (cortisol, DHEA, and CgA) and to evaluate the immunopathogenesis of Th17.

The findings of this study may significantly contribute to clinical practice regarding the early diagnosis and management of periodontal disease in individuals with psoriasis. It also aims to encourage multidisciplinary approaches by providing a holistic understanding of the effects of stress on the immune system and periodontal health.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 65
* Being diagnosed with psoriasis by a dermatologist
* Having at least 20 teeth
* Not having received periodontal treatment in the last 6 months
* Not having taken antibiotics, steroids, and/or nonsteroidal anti-inflammatory drugs in the last 3 weeks
* Not having any autoimmune disease, osteoporosis, or cancer
* Not using immunosuppressive drugs, oral contraceptives, or bisphosphonates
* Not being pregnant
* Not having an active infectious disease (acute hepatitis, tuberculosis, AIDS)
* Not using chronic medications that affect periodontal tissues (cyclosporine A, phenytoin)
* Not having taken antioxidant supplements in the last 6 months

Exclusion Criteria:

* <20 teeth
* Any significant oral infection (i.e., herpes or candidiasis)
* Oral injuries or bleeding unrelated to periodontitis
* Periodontal therapy and antibiotic therapy within the past 3 months
* Salivary gland dysfunction
* Acute illness (fever, sore throat)
* Systemic illness, mental illness, immunosuppressive drugs or immunodeficiency
* Pregnancy or breastfeeding
* Use of antidepressants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with psoriasis who came to the Periodontology Clinic of Recep Tayyip Erdoğan University Faculty of Dentistry for routine periodontal treatment
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-04-06 (Estimated)

PRIMARY OUTCOMES:
Gingival Crevicular Fluid (GCF) Collection | Day 1
  Specimens will be collected from four different teeth from each participant, each with the deepest pocket. Before collection, supragingival plaque will be gently removed with sterile curettes, the surfaces will be dried, and the tissue will be isolated with cotton rolls. Filter paper strips will be carefully inserted into the sulcus until slight resistance is felt, or no deeper than 1 mm to prevent mechanical trauma in patients with periodontitis. The strips will be left in the sulcus/pocket for 30 seconds. The GCF volume of each strip will be measured using a pre-calibrated electronic device (Peritron 8000). Four strips from each participant will be placed in coded sterile Eppendorf tubes and stored at -80°C until analysis.
Saliva sampling | Day 1
  Prior to saliva collection, participants will be instructed to abstain from caffeine and/or nicotine for at least 4 hours and alcohol for at least 24 hours. Participants will be asked to rinse their mouth with water and wait 5 minutes to prevent contamination. After waiting, they will be asked to collect saliva in the bottom of their mouth and then spit into a sterile metal cup for another 5 minutes. Unstimulated saliva samples will be transferred to sterile Eppendorf tubes. Saliva flow rate will be calculated by dividing the total saliva volume by the collection time for each participant. Samples will be stored at -80°C until the day of laboratory analysis.
Clinical Periodontal Parameters (Plaque Index) | Day 1
  Plaque Index (PI) (Silness and Löe, 1964) This index is used to evaluate the amount of dental plaque accumulation on tooth surfaces. Each tooth's four surfaces (buccal, lingual, mesial, distal) are examined using a probe or visually. Each surface is scored from 0 to 3. The average score is calculated for each tooth. The overall plaque index is obtained by averaging the scores from all examined teeth.
  Score Description 0 No plaque.
  1. No visible plaque, but a slight film of plaque is detected when a probe is run along the gingival margin.
  2. Visible plaque along the gingival margin, forming a continuous band.
  3. Abundant plaque covering the gingival area and extending toward the middle of the tooth surface, including the interproximal spaces.
Clinical Periodontal Parameters (Gingival Index) | Day 1
  The Gingival Index is used to assess the presence and severity of gingival inflammation (gingivitis).
  Four surfaces of each tooth (buccal, lingual, mesial, distal) are examined visually and with a periodontal probe. The evaluation considers color changes, edema (swelling), tissue consistency, and bleeding on probing. Each surface is scored from 0 to 3.
  The average score per tooth is calculated, and then the overall average is used to determine the individual's GI score.
  Score Description 0 Healthy gingiva: normal color and texture, no bleeding
  1. Mild inflammation: slight color change and swelling, no bleeding on probing
  2. Moderate inflammation: redness, edema, soft tissue, bleeding on probing
  3. Severe inflammation: marked redness and swelling, ulceration, possible spontaneous bleeding
Periodontal Clinical Parametres (Bleeding on Probing Index) | Day 1
  This index is used to assess the presence and severity of gingival inflammation by observing bleeding after gentle pressure is applied to the gingival sulcus using a periodontal probe. A thin periodontal probe is gently inserted into the gingival sulcus with light pressure (approximately 20-25 grams). Bleeding occurring within 10-30 seconds is observed. Each measurement site is recorded as either "bleeding present" or "bleeding absent." Presence of bleeding is an early and sensitive indicator of gingival inflammation.
  Score Description:
  0 No bleeding
  1 Bleeding present (mild or severe)
Periodontal Clinical Parametres (Probing Pocket Depth) | Day 1
  Using a Williams periodontal probe, the distance between the gingival margin and the base of the periodontal pocket is measured in millimeters at six sites per tooth: mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual. All teeth are measured. The values obtained from each site are summed and then divided by the total number of sites measured. This gives the average probing depth for the individual.
  Measurement Interpretation 1-3 mm Healthy sulcus 4-5 mm Shallow to moderate pocket
  ≥6 mm Deep periodontal pocket (advanced disease)
Periodontal Clinical Parametres (Clinical Attachment Loss) | Day 1
  Using a Williams periodontal probe, the distance between the enamel-cementum junction and the base of the periodontal pocket is measured in millimeters at six sites per tooth: mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual. All teeth are measured. The values obtained from each site are summed and then divided by the total number of sites measured. This gives the average probing depth for the individual.
  CAL Value Interpretation 0-1 mm Healthy / minimal loss 2-3 mm Mild attachment loss 4-5 mm Moderate attachment loss
  ≥6 mm Severe attachment loss
Application of the Social Appearance Anxiety Scale | Day 1
  This 16-item scale concerns how patients feel about their appearance. Each item is scored from 1 to 5 as follows: 1, strongly disagree; 2, somewhat disagree; 3, unsure; 4, somewhat agree; and 5, strongly agree. Scores range from 16 to 80, with higher scores representing greater social appearance anxiety.

SECONDARY OUTCOMES:
Analysis of cortisol, dehidroepiandrosteron (DHEA) and chromogranin A | 5th month
  Salivary cortisol, DHEA, and chromogranin A will be obtained from unstimulated whole saliva samples. Human salivary cortisol will be measured using a commercial enzyme-linked immunosorbent assay (ELISA) radioenzyme immunoassay kit according to the manufacturer's instructions. An ELISA kit will be used to measure DHEA, and the Human Chromogranin A ELISA Kit will be used to measure chromogranin A levels. Saliva samples will be kept on ice and stored at -20°C until analyzed. On the day of analysis, saliva samples will be centrifuged at 2000×g for 10 minutes to remove particulate material. All samples will be processed in triplicate during the same assay. Statistical analyses will be performed using the average of three replicate measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontology of the Faculty of Dentistry of Recep Tayyip Erdogan University, Rize, Rize Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No